CLINICAL TRIAL: NCT01054664
Title: The Incidence of Occult Hepatitis C Virus Infection in Hemodialysed Patients With Liver Enzymes Disturbances
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Plotkin Eleonora, Clalit Health services
Other Study IDs: nephrop003
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2010-01

CONDITIONS: Hemodialysed Patients With Impaired Liver Enzymes
Keywords: liver enzymes; peripheral mononuclear blood cells; hemodialysis; hepatitis C; RNA
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- impaired liver enzymes
- normal liver enzymes
- hepatitis C antibodies positive

SUMMARY:
To assess the incidence of occult hepatitis C virus in hemodialysed patients with mild impairment of liver enzymes

DETAILED DESCRIPTION:
occult hepatitis C virus will be checked in monocytes of hemodialyzed patients with permanent mild impairment of liver enzymes This population has no evidence of hepatitis B or C according to standard laboratory tests (HVC antibodies,HCV PCR, hepatitis B antibodies) Hepatitis C virus RNA will be performed in peripheral blood mononuclear cells of hemodialysed patients

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysed patients with impaired liver enzymes

Exclusion Criteria:

* hepatitis B and C positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hemodialysis patients with impaired liver enzymes
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-02

CONTACTS AND LOCATIONS:
Locations (1):
- Plotkin Eleonora, Kfar Saba, Israel